CLINICAL TRIAL: NCT04172779
Title: Phase II Clinical Trial of Low-dose Erlotinib for Hepatocellular Carcinoma Chemoprevention
Brief Title: Erlotinib for Hepatocellular Carcinoma Chemoprevention
Acronym: ECHO-B
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Yujin Hoshida, MD, PhD, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU-2019-1515; P50CA295495 (NIH)
Record Dates: First submitted 2019-11-17; First posted 2019-11-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cirrhosis, Liver; Advanced Liver Fibrosis
Keywords: hepatocellular carcinoma; chemoprevention
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Erlotinib treatment (Experimental)
  Interventions: Drug: erlotinib hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: erlotinib hydrochloride — Oral administration of erlotinib 50mg (two 25mg capsules)
  Arms: Erlotinib treatment
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This phase II randomized placebo-controlled trial studies low-dose erlotinib treatment to assess its efficacy and safety to prevent development of hepatocellular carcinoma in patients with advanced liver fibrosis or cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years-old)
* Clinically and/or histologically diagnosed advanced liver fibrosis or cirrhosis
* No active hepatic decompensation
* No prior history of HCC
* FIB-4 index > 3.25
* PLSec score ≥ 3
* Adequate hematologic, hepatic, and renal function, Karnofsky performance status score ≥70
* Both sexes and all racial/ethnic groups will be considered

Exclusion Criteria:

* Prior treatment with epidermal growth factor receptor (EGFR) inhibitors
* Uncontrolled intercurrent, use of CYP3A4 modulators
* Erlotinib treatment <4 weeks or <80% of planned regimen at the end of week 4
* HCC development during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Modulation of serum protein signature associated with hepatocellular carcinoma (HCC) risk | Baseline, 24 weeks
  The relationship between the treatment and modulation of a serum protein signature associated with HCC risk (PLSec) will be assessed. PLSec-based HCC risk level (i.e., PLSec score) will be compared between baseline and at the end of treatment, and magnitude of the modulation will be measured as delta-PLSec and compared between the treatment groups by t-test and Wilcoxon rank-sum test.

SECONDARY OUTCOMES:
Overall adverse event profile for erlotinib hydrochloride | Baseline, 24 weeks
  Graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5. The maximum grade for each type of adverse event will be recorded for each participant and frequency tables will be reviewed to determine the overall patterns. The number and severity of adverse events will be tabulated and summarized across all grades. Grade 3+ adverse events will be similarly described and summarized separately. Overall toxicity incidence, as well as toxicity profiles will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Change in quality of life (QOL) | Baseline, 24 weeks
  QOL will be measured by using Chronic Liver Disease Questionnaire (CLDQ), and compared between baseline and end of the treatment. Frequency distributions, graphical techniques and other descriptive measures will be used to summarize the results. Paired t-test will be used to assess change of the measurements.

OTHER OUTCOMES:
Molecular tissue transcriptome signature associated with HCC risk | Baseline, 24 weeks
  When optional liver biopsy tissues are obtained, the relationship between the treatment and modulation of a gene expression signature associated with HCC risk will be assessed. Expression levels of the signature genes will be compared between baseline and at the end of treatment, and magnitude of the modulation will be measured by Kolmogorov-Smirnov statistic-based Combined Enrichment Score (CES) and tested by t-test and Wilcoxon rank-sum test.
Changes in phospho-ERK levels in the liver | Baseline, 24 weeks
  When optional liver biopsy tissues are obtained, the relationship between dose-level and staining of biomarkers in the liver will be assessed. The baseline biomarker expression levels across all the dose levels using analysis of variance (ANOVA) or the nonparametric equivalent will be compared. The changes in these biomarker values will be assessed using the Wilcoxon signed-rank test and compare these changes across dose levels using ANOVA. Graphical methods will be used to assess the differences in these biomarker values across dose levels. All categorical variables will be analyzed using chi-square or Fisher's exact tests.
Changes in PCNA levels in the liver | Baseline, 24 weeks
  When optional liver biopsy tissues are obtained, the relationship between dose-level and staining of biomarkers in the liver will be assessed. The baseline biomarker expression levels across all the dose levels using ANOVA or the nonparametric equivalent will be compared. The changes in these biomarker values will be assessed using the Wilcoxon signed-rank test and compare these changes across dose levels using ANOVA. Graphical methods will be used to assess the differences in these biomarker values across dose levels. All categorical variables will be analyzed using chi-square or Fisher's exact tests.
Changes in EGF levels in the liver | Baseline, 24 weeks
  When optional liver biopsy tissues are obtained, the relationship between dose-level and staining of biomarkers in the liver will be assessed. The baseline biomarker expression levels across all the dose levels using ANOVA or the nonparametric equivalent will be compared. The changes in these biomarker values will be assessed using the Wilcoxon signed-rank test and compare these changes across dose levels using ANOVA. Graphical methods will be used to assess the differences in these biomarker values across dose levels. All categorical variables will be analyzed using chi-square or Fisher's exact tests.
Changes in alphaSMA levels in the liver | Baseline, 24 weeks
  When optional liver biopsy tissues are obtained, the relationship between dose-level and staining of biomarkers in the liver will be assessed. The baseline biomarker expression levels across all the dose levels using ANOVA or the nonparametric equivalent will be compared. The changes in these biomarker values will be assessed using the Wilcoxon signed-rank test and compare these changes across dose levels using ANOVA. Graphical methods will be used to assess the differences in these biomarker values across dose levels. All categorical variables will be analyzed using chi-square or Fisher's exact tests.
Changes in GSTp levels in the liver | Baseline, 24 weeks
  When optional liver biopsy tissues are obtained, the relationship between dose-level and staining of biomarkers in the liver will be assessed. The baseline biomarker expression levels across all the dose levels using ANOVA or the nonparametric equivalent will be compared. The changes in these biomarker values will be assessed using the Wilcoxon signed-rank test and compare these changes across dose levels using ANOVA. Graphical methods will be used to assess the differences in these biomarker values across dose levels. All categorical variables will be analyzed using chi-square or Fisher's exact tests.
Liver stiffness measurement by transient elastography | Baseline, 24 weeks
  The change in liver stiffness measurement (LSM) by transient elastography will be evaluated by comparing baseline and at the end of the treatment and compared between the treatment groups by t-test and Wilcoxon rank-sum test.
HCC incidence | through study completion, an average of 3 year
  HCC incidence after completing the planned treatment will be recorded via standard-care semi-annual HCC screening with ultrasound and AFP. The association of the treatment and HCC incidence will be assessed by Kaplan-Meier method, log-rank test, and Cox regression. Correlation with the primary endpoint will also be assessed. The semi-annual HCC screening will be continued indefinitely and the correlation analysis will be continued.

CONTACTS AND LOCATIONS:
Overall Officials: Yujin Hoshida, Principal Investigator — UT Southwestern; Amit Singal, MD, MS, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.